CLINICAL TRIAL: NCT01182441
Title: Prospective Randomized Evaluation of the WATCHMAN LAA Closure Device in Patients With Atrial Fibrillation (AF) Versus Long Term Warfarin Therapy
Brief Title: Evaluation of the WATCHMAN Left Atrial Appendage (LAA) Closure Device in Patients With Atrial Fibrillation Versus Long Term Warfarin Therapy
Acronym: PREVAIL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT1004
Record Dates: First submitted 2010-08-12; First posted 2010-08-16 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2017-03

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: atrial fibrillation; stroke; TIA; trans ischemic attack; warfarin; Coumadin
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WATCHMAN (Experimental): Subjects assigned to receive the WATCHMAN device.
  Interventions: Device: WATCHMAN Device
- Warfarin (Active Comparator): Subjects assigned to warfarin therapy.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Device: WATCHMAN Device — WATCHMAN Left Atrial Appendage Closure Technology
  Arms: WATCHMAN
Drug: Warfarin — Warfarin dosage prescribed by study physician to adequately maintain an INR of 2.0-3.0
  Other Names: Coumadin
  Arms: Warfarin

SUMMARY:
This was a prospective, randomized, multicenter study to provide additional information on the safety and efficacy of the WATCHMAN LAA Closure Technology. The purpose of the PREVAIL study was to confirm the efficacy endpoint as demonstrated in the PROTECT AF pivotal study and to further demonstrate that the WATCHMAN LAA Closure Technology is safe and effective in subjects with non-valvular atrial fibrillation who require anticoagulation therapy for potential thrombus formation.

ELIGIBILITY:
Key Inclusion Criteria:

* Paroxysmal, persistent or permanent non-valvular AF
* Eligible for long-term warfarin therapy
* Eligible to come off warfarin therapy
* Calculated CHADS2 score of 2 or greater. Also patients with a CHADS2 score of 1 may be included if any of the following apply:

  * Female age 75 or older
  * Baseline LVEF ≥ 30 and < 35%
  * Aged 65-74 and has diabetes or coronary artery disease
  * Aged 65 or greater and has congestive heart failure

Key Exclusion Criteria:

* Contraindicated/allergic to aspirin
* Indicated for clopidogrel therapy or has taken clopidogrel within 7 days prior to enrollment
* History of atrial septal repair or has an ASD/PFO device
* Implanted mechanical valve prosthesis
* NYHA Class IV CHF
* Resting heart rate > 110 bpm
* Participated previously in the PROTECT AF or CAP Registry studies

Key Echo Exclusion Criteria:

* LVEF < 30%
* Existing pericardial effusion > 2mm
* High risk PFO
* Significant mitral valve stenosis
* Complex atheroma with mobile plaque of the descending aorta and/or aortic arch
* Cardiac tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Holmes, M.D., Principal Investigator — Mayo Clinic; Vivek Y. Reddy, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (41):
- United States (41):
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Arizona Heart Rhythm Research Center, Scottsdale, Arizona
  - Foundation for Cardiovascular Medicine, La Jolla, California
  - Scripps Green, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Orange County Heart, Orange, California
  - St. John's Hospital / Pacific Heart, Santa Monica, California
  - Zasa Clinical Research, Atlantis, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - North Shore University, Evanston, Illinois
  - Iowa Heart Center, Des Moines, Iowa
  - Central Baptist Hospital, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - William Beaumont, Royal Oak, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Cardiology Associates of N. Mississippi, Tupelo, Mississippi
  - St. Luke's Hospital, Kansas City, Missouri
  - St. John's Mercy, St Louis, Missouri
  - Bryan LGH, Lincoln, Nebraska
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - New York University Medical Center, New York, New York
  - Mt. Sinai School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Lindner Clinical Trial Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Moffitt Heart & Vascular, Wormleysburg, Pennsylvania
  - St. Thomas Research Institute, Nashville, Tennessee
  - Texas Cardiac Arrhythmia, Austin, Texas
  - Baylor Research Institute, Dallas, Texas
  - Methodist Hospital, Houston, Texas
  - Intermountain Medical Center, Salt Lake City, Utah
  - Fletcher Allen, Burlington, Vermont
  - Swedish Medical Center, Seattle, Washington
  - St. Luke's Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dukkipati SR, Holmes DR Jr, Doshi SK, Kar S, Singh SM, Gibson D, Price MJ, Natale A, Mansour M, Sievert H, Houle VM, Allocco DJ, Reddy VY. Impact of Peridevice Leak on 5-Year Outcomes After Left Atrial Appendage Closure. J Am Coll Cardiol. 2022 Aug 2;80(5):469-483. doi: 10.1016/j.jacc.2022.04.062. PMID 35902169
- [Derived] Friedman DJ, Du C, Wang Y, Agarwal V, Varosy PD, Masoudi FA, Holmes DR, Reddy VY, Price MJ, Curtis JP, Freeman JV. Patient-Level Analysis of Watchman Left Atrial Appendage Occlusion in Practice Versus Clinical Trials. JACC Cardiovasc Interv. 2022 May 9;15(9):950-961. doi: 10.1016/j.jcin.2022.02.029. PMID 35512918
- [Derived] Brouwer TF, Whang W, Kuroki K, Halperin JL, Reddy VY. Net Clinical Benefit of Left Atrial Appendage Closure Versus Warfarin in Patients With Atrial Fibrillation: A Pooled Analysis of the Randomized PROTECT-AF and PREVAIL Studies. J Am Heart Assoc. 2019 Dec 3;8(23):e013525. doi: 10.1161/JAHA.119.013525. Epub 2019 Nov 22. PMID 31752643
- [Derived] Price MJ, Reddy VY, Valderrabano M, Halperin JL, Gibson DN, Gordon N, Huber KC, Holmes DR Jr. Bleeding Outcomes After Left Atrial Appendage Closure Compared With Long-Term Warfarin: A Pooled, Patient-Level Analysis of the WATCHMAN Randomized Trial Experience. JACC Cardiovasc Interv. 2015 Dec 28;8(15):1925-1932. doi: 10.1016/j.jcin.2015.08.035. Epub 2015 Nov 25. PMID 26627989

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | WATCHMAN | Warfarin
Started | 269 | 138
Completed | 49 | 19
Not Completed | 220 | 119
Not completed — Patient Still in Follow-up | 152 | 72
Not completed — Death | 37 | 25
Not completed — Implant Attempt Unsuccessful | 13 | 0
Not completed — Lost to Follow-up | 5 | 8
Not completed — Withdrawal by Subject | 6 | 13
Not completed — Implant Not Attempted | 4 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | WATCHMAN | Warfarin | Total
Number analyzed (Participants) | 269 | 138 | 407
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.0 (7.4) | 74.9 (7.2) | 74.3 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 35 | 122
  Male | 182 | 103 | 285
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2
  Black/Aftrican American | 6 | 1 | 7
  Caucasian | 253 | 131 | 384
  Hispanic/Latino | 6 | 5 | 11
  Native American Indian/Alaskan Native | 1 | 0 | 1
  Other | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 269 | 138 | 407
CHADS2 Stroke Risk Score [Mean (Standard Deviation); unit: scores on a scale] — The CHADS2 score is used to estimate the risk of stroke in patients with non-rheumatic atrial fibrillation. To calculate the CHADS2 score, one point was assigned each for the presence of Congestive heart failure, history of Hypertension, Age 75 years or older, and Diabetes, and two points assigned for prior Stroke or TIA.
  The range for this stroke scale is 0, with an annual stroke risk of 1.9%, to 6, which represents the highest risk of stroke for these patients using this scale and an annual stroke risk of 18.2% (JAMA. 285 (22): 2864-70).
  scores on a scale | 2.6 (1.0) | 2.6 (1.0) | 2.6 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint (Device Group Only)
Description: 7-Day procedure rate of death, ischemic stroke, systemic embolism and complications requiring major cardiovascular or endovascular intervention.
Time Frame: 7-Day
Measure: Count of Participants; unit: Participants
Arm/Group | WATCHMAN
Number analyzed (Participants) | 269
Participants | 6
Statistical Analysis 1: Comparison: WATCHMAN; Bayesian calculations were used to incorporate the data from PROTECT AF CAP Registry through a conjugate beta-binomial model. A one-sided upper 95% credible interval for the event rate was calculated based off this posterior distribution; Test type: Superiority — Success for this endpoint was achieved if the probability of experiencing an event was statistically less than the performance goal, defined as 2.67%, with an upper bound of the one-sided 95% credible interval less than the performance goal; probability of experiencing an event = 2.2, 95% CI 1-sided [upper limit 2.652]

2. Primary Outcome: Composite of Stroke, Systemic Embolism, and Death (Cardiovascular and Unknown)
Description: The endpoint was analyzed using a Bayesian piecewise exponential model with the historical priors based on data from the previous pivotal study PROTECT AF. This was a non-inferiority design with comparison of rate ratio of 18-month event rates of the Device and Control groups. The 18-month rate represents the probability of an event occurring within 18 months, and the 18-month rate ratio is a mean of the rate ratios. The primary endpoint was based on a calculation of the probability of events at 18 months but the statistical piecewise hazards model does not require the observation of any subjects out to 18-months.
Time Frame: 18 month rate
Measure: Number; unit: Probability of events within 18 months
Arm/Group | WATCHMAN | Warfarin
Number analyzed (Participants) | 269 | 138
Probability of events within 18 months | 0.064 | 0.063
Statistical Analysis 1: Comparison: WATCHMAN vs Warfarin; A Bayesian piecewise exponential model was used to model the 18-month event rates. Historical priors for each interval model were based on PROTECT AF. Hazards were modeled for 0-7 day, 7-60 day, 60-182 day, and 182+ day intervals. Event rates were estimated separately by treatment group and event type. The posterior distribution for the 18-month event rate ratio (WATCHMAN vs. Warfarin), and the corresponding equitailed 95% credible interval, were determined via Monte Carlo simulations; Test type: Non-Inferiority — This endpoint is met if the 95% Credible Interval for the rate ratio of WATCHMAN versus Warfarin is entirely less than 1.75; Risk Ratio (RR) = 1.07, 95% CI 2-sided [0.57 to 1.89]

3. Primary Outcome: Composite of Ischemic Stroke or Systemic Embolism
Description: Composite of ischemic stroke or systemic embolism excluding events that occurred in the first 7 days following randomization
Time Frame: Day 8 to 18-months
Measure: Number; unit: Probability of events within 18-months
Arm/Group | WATCHMAN | Warfarin
Number analyzed (Participants) | 269 | 138
Probability of events within 18-months | 0.0253 | 0.0200
Statistical Analysis 1: Comparison: WATCHMAN vs Warfarin; A Bayesian piecewise exponential model was used to model the 18-month event rates. Historical priors for each interval were based on PROTECT AF. Hazards were modeled for 0-7 day, 7-60 day, 60-182 day, and 182+ day intervals. Event rates were estimated separately for the WATCHMAN and Warfarin groups. The posterior distribution for the 18-month event rate ratio (WATCHMAN vs. Warfarin), and the corresponding equitailed 95% credible interval, were determined via Monte Carlo simulations; Test type: Non-Inferiority — This endpoint is met if either the 95% Credible Interval for the risk ratio < 2.0 or the 95% Credible Interval for the risk difference is < 0.0275; Risk Difference (RD) = 0.0053, 95% CI 2-sided [-0.0190 to 0.0273]
Statistical Analysis 2: Comparison: WATCHMAN vs Warfarin; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Risk Ratio (RR) = 1.6, 95% CI 2-sided [0.5 to 4.2]

ADVERSE EVENTS:
Time Frame: Randomization through 5-years
Arm/Group | WATCHMAN | Warfarin
All-Cause Mortality (participants affected / at risk) | 37/269 | 25/138
Serious Adverse Events (participants affected / at risk) | 86/269 | 44/138
Other Adverse Events (participants affected / at risk) | 38/269 | 10/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WATCHMAN (N=269) | Warfarin (N=138)
AV fistula (Vascular disorders) | 1 (1) | 0 (0)
Anemia requiring transfusion (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Bleeding, other (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Cardiac perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cranial bleed (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 36 (36) | 24 (24)
Device embolization (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Device thrombus (General disorders) | 1 (1) | 0 (0)
Epistaxis (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Gastrointestinal bleeding (Gastrointestinal disorders) | 19 (19) | 12 (12)
Hematoma (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Hematuria (Gastrointestinal disorders) | 1 (1) | 2 (2)
Infection (Infections and infestations) | 3 (3) | 0 (0)
Major bleeding requiring transfusion (Blood and lymphatic system disorders) | 6 (6) | 2 (2)
Other study related (General disorders) | 6 (7) | 1 (1)
Pericardial effusion with cardiac tamponade (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Pseudoaneurysm (Vascular disorders) | 1 (1) | 0 (0)
Rectal bleeding (Gastrointestinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hemorrhagic stroke (Cardiac disorders) | 2 (2) | 3 (3)
Ischemic stroke (Cardiac disorders) | 15 (16) | 4 (4)
Subdural hematoma (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Systemic embolism (Cardiac disorders) | 1 (1) | 0 (0)
Transient ischemic attack (Cardiac disorders) | 5 (6) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WATCHMAN (N=269) | Warfarin (N=138)
Anemia requiring transfusion (Blood and lymphatic system disorders) | 4 (5) | 0 (0)
Bleeding, other (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Device thrombus (General disorders) | 15 (16) | 0 (0)
Epistaxis (Ear and labyrinth disorders) | 5 (5) | 1 (2)
Gastrointestinal bleeding (Gastrointestinal disorders) | 2 (2) | 2 (3)
Hematuria (Gastrointestinal disorders) | 1 (1) | 3 (3)
Oral bleeding (General disorders) | 2 (2) | 0 (0)
Other study related (General disorders) | 2 (2) | 0 (0)
Pericardial effusion, non-serious (Cardiac disorders) | 2 (2) | 0 (0)
Pseudoaneurysm (Vascular disorders) | 2 (2) | 0 (0)
Rectal bleeding (Gastrointestinal disorders) | 2 (2) | 0 (0)
Transient ischemic attack (Cardiac disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No